CLINICAL TRIAL: NCT04721340
Title: Upper Limb Assessment in Multiple Sclerosis: The Minnesota Manual Dexterity Test As A Measure Of Hand Function
Brief Title: The Minnesota Manual Dexterity Test As A Measure Of Hand Function in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Uğur OVACIK, Lecturer in physiotherapy and principal investigator of the study, Istanbul Aydın University
Other Study IDs: 2020/03
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; upper limb; manual dexterity; assessment; minnesota manual dexterity test
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: people with multiple sclerosis
  Interventions: Other: Test Group
- Control Group: healthy volunteers
  Interventions: Other: Control Grup

INTERVENTIONS:
Other: Test Group — Individuals who meet the inclusion criteria will be evaluated for manual dexterity, performance, muscle strength and fatigue, respectively, on a predetermined day.
  Groups: Test Group
Other: Control Grup — Individuals who meet the inclusion criteria will be evaluated for manual dexterity, performance, muscle strength and fatigue, respectively, on a predetermined day.
  Groups: Control Group

SUMMARY:
The aim of the study is to report the results of manual dexterity using the Minnesota Manual Dexterity Test in people with Multiple Sclerosis.

DETAILED DESCRIPTION:
Upper limb can be affected even in early stage in people with Multiple Sclerosis (pwMS). Manual dexterity is important to maintain upper limb function and 9-Hole Peg Test (9HPT) is used as gold standard to assess dexterity in pwMS. There are no studies evaluating manual dexterity with the Minnesota Manual Dexterity Test (MMDT) in pwMS. This study aims to:

1. reporting the results of manual dexterity using the Minnesota Manual Dexterity Test and comparing the test results with healthy volunteers,
2. examining the relationship between MMDT and 9HPT, ABILHAND, grip strength, pinch strength, fatigue.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 18-65;
* (2) definitive diagnosis of MS according to McDonald criteria;
* (3) ability to read and write in Turkish.

Exclusion Criteria:

* (1) acute attacks of MS (within 3 months);
* (2) cognitive impairment (Mini Mental test result 24 points and below);
* (3) having spasticity (3 and above according to Modified Ashworth Scale)
* (4) any chronic disease other than MS;
* (5) being addicted to alcohol or drugs,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Test group: 80 people with multiple sclerosis will be evaluated. Inclusion and exlusion criteria listed above. Control group: 40 healthy volunteers with demographic characteristics similar to people with multiple sclerosis will be evaluated to compare people with multiple sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-16 (Actual)

PRIMARY OUTCOMES:
Minnesota Manual Dexterity Test | baseline (on the predetermined assessment day)
  to assess manual dexterity, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
9-Hole Peg Test | baseline (on the predetermined assessment day)
  to assess manual dexterity. higher scores mean a worse outcome.
ABILHAND | baseline (on the predetermined assessment day)
  to assess for performance of activity. score range 0-46 point, higher scores mean a better outcome.
grip strength | baseline (on the predetermined assessment day)
  using hand dynamometer. higher scores mean a better outcome.
pinch strength | baseline (on the predetermined assessment day)
  using pinchmeter. higher scores mean a better outcome.
Fatigue Severity Scale | baseline (on the predetermined assessment day)
  to assess fatigue. score range 0-7 point, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Küçükçekmece, Turkey (Türkiye)